CLINICAL TRIAL: NCT03032367
Title: TASK-002: Bioequivalence of Bedaquiline 400mg Administered in Crushed Form Compared to Tablet Form in Healthy Male and Female Adults Under Fed Conditions (BDQ Crush Study)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: US National Institute of Allergy and Infectious Diseases (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TASK-002
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — bedaquiline

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive study drug (bedaquiline (BDQ)) in either tablet form or crushed form in one of two sequences:
  Sequence 1: BDQ 4 x 100mg administered in a whole tablet form, followed by BDQ 4 x 100mg administered in crushed form as a once only dose
  Sequence 2: BDQ 4 x 100mg administered in crushed form, followed by BDQ 4 x 100mg administered in tablet form as a once only dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (Other): Bedaquiline 4 x 100mg administered in a whole tablet form, followed by bedaquiline 4 x 100mg administered in crushed form as a once only oral dose
  Interventions: Drug: bedaquiline
- Sequence 2 (Other): Bedaquiline 4x 100mg administered in crushed form, followed by bedaquiline 4 x 100mg administered in a whole tablet form, as a once only oral dose
  Interventions: Drug: bedaquiline

INTERVENTIONS:
Drug: bedaquiline
  Other Names: Sirturo

SUMMARY:
This is a randomized, open-label, cross-over study comparing the bioequivalence of bedaquiline administered in whole tablet form versus bedaquiline administered in crushed (experimental) form in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a randomized, open-label, cross-over, bioequivalence study with two single treatment periods, separated by a 14-day wash-out period, conducted among 24 healthy adult males and females, who receive 400mg (4 x 100mg) bedaquiline orally in one of two sequences: either first in whole tablet form and second in crushed (experimental) form, or vice versa under fed conditions. The bioequivalence evaluation will be based on primary pharmacokinetic (pk) parameters affecting the extent of absorption, i.e., the bioavailability. If bioequivalence is not shown, the knowledge about the differences in bioavailability between whole and crushed tablets will be used for assessing the need of dose adjustment in children receiving the crushed form.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, including HIV testing
* Male or female between 18 and 55 years of age inclusive
* Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive
* In the opinion of the investigator, able to comply with the requirements of the protocol e.g. able to attend all visits for PK analysis
* Be of non-childbearing potential or using effective methods of birth control

Exclusion Criteria:

* Known or suspected hypersensitivity or intolerance to bedaquiline or any other constituents of the study drug, i.e. lactose
* A history or clinical evidence of any clinically significant cardiac condition including but not limited to congenital long QT syndrome, Torsades de Pointes, bradyarrhythmias
* Uncontrolled cardiac dysrhythmias
* Severe hepatic impairment (Child Pugh C)
* History, symptoms or signs of heart failure
* History, symptoms or signs of hypothyroidism, whether currently controlled or uncontrolled
* Any other serious uncontrolled medical condition or clinically significant abnormality, which, in the opinion of the investigator, might compromise the safety of the subject or which might interfere with the study.
* Evidence of clinically significant (as judged by the investigator), metabolic, gastrointestinal, cardiovascular, musculoskeletal, ophthalmological, pulmonary, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities.
* Concomitant use of medicines known to prolong the QTc interval, or use of CYP3A4 inducers/inhibitors including but not limited to, carbamazepine, phenytoin, St. John's wort, ciprofloxacin, erythromycin, clarithromycin, fluconazole, ketoconazole, ritonavir or other anti-retroviral medications, fluoroquinolones and clofazamine.
* HIV positive, already known or as per HIV test done at screening.
* Hepatitis B or C positive
* QTc prolongation as per ECG with a QTcF of >450msec or any other significant finding on the ECG as per the investigator
* Receipt of any study drug within the past 3 months.
* Scheduled to receive any other investigational drug during the course of the study.
* Known or suspected, current or history of within the past 2 years, alcohol or drug abuse, that is, in the opinion of the Investigator, sufficient to compromise the safety or cooperation of the volunteer.
* Evidence or suspicion of active TB or documented recent (within the last year) household contact with an infectious TB case.
* The following toxicities at screening as defined by the DAIDS toxicity table (November 2014)

  1. aspartate aminotransferase (AST) grade 3 (≥3.0 x ULN)
  2. alanine aminotransferase (ALT) grade 3 (≥3.0 x ULN)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2017-01-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence of bedaquiline 4 x 100mg given to healthy adult males and females orally in tablet form compared to crushed form | Two single treatment sequences, separated by a 14-day wash-out period
  The bioequivalence evaluation will be based on primary PK parameters affecting the extent of absorption, i.e. the bioavailability.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannine du Bois, MD, Study Chair — TASK Clinical Research Centre; Anthony Garcia-Pratts, MD, Study Chair — Desmond Tutu TB Centre, Stellenbosch University
Locations (1):
- TASK Clinical Research Centre, Bellville, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No